CLINICAL TRIAL: NCT01993966
Title: Mechanism of (-)-Epigallocatechin -3-gallate (EGCG) to Modulate the Cytotoxic Effects of Chemotherapeutic Agents in Human Urothelial Carcinoma Cells
Brief Title: EGCG Modulate the Cytotoxic Effects of Chemotherapeutic Agents in Human Urothelial Carcinoma Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201308047RIN; 103-002509 (Other Grant/Funding Number: National Taiwan University Hospital)
Record Dates: First submitted 2013-10-24; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial carcinoma (UC),; (-)-epigallocatechin-3-gallate(EGCG),; chemotherapy,; cytotoxicity,; drug resistance,; xenograft.
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- drug-resistant: specimens com from drug-resistant bladder urothelial carcinoma patients
- normal: specimens come from normal bladder urothelial carcinoma patients
- non-tumoral: specimens come from non-tumoral patients

SUMMARY:
Urothelial carcinoma (UC) is the most common cancer of urinary tract. Patients with metastatic UC are usually treated with systemic chemotherapy. There still existed 30% to 50% of advanced UC not responsive to cisplatin-based chemotherapy; the prognosis for patients with metastatic UC remains poor.

DETAILED DESCRIPTION:
(-)-epigallocatechin -3-gallate (EGCG) is the most abundant polyphenol compound from green tea, representing ~16.5% of the water-extractable fraction. EGCG have various bioactivities and can bind and regulate a wide range of molecular involved in cell cycle, signal transduction, and protein degradation. However, the anticancer effects of EGCG on UC have not been thoroughly explored. Our preliminary data show that EGCG alone can inhibit cell proliferation and induce apoptosis with the activation of caspases and PARP in a time dependent manner. Moreover, EGCG can enhance the cytotoxicity of several chemotherapeutic drugs in vitro. The underlying mechanism seems to be associated with Akt and ERK pathway. We will also check the Akt and ERK protein level by immunohistochemical staining in clinically chemoreistant bladder urothelial carcinoma specimens to further prove our in vitro findings. We will further confirm the effect of chemotherapeutic drugs combined with EGCG on UC in vivo via xenograft model.

The specific aims of the study are:

1. To explore the anti-tumor effects of EGCG on human UC cells and elucidate the possible mechanisms.
2. To study the combinative cytotoxic effect of EGCG with other chemotherapeutic agents such as cisplatin, doxorubicin and gemcitabine on UC cells; moreover, to investigate the underlying mechanisms.
3. To investigate the expression level of phospho-Akt and phospho-ERK in clinically chemoreistant bladder urothelial carcinoma specimens to further confirm our finding in clinical events. .
4. To prove the in vitro findings and confirm the combinative efficacy of EGCG with chemotherapeutic agents in vivo by using the xenograft animal model.
5. To establish a novel therapeutic strategy for treatment of UC.

ELIGIBILITY:
Inclusion Criteria:

* In January 2008 to December 2012 at the National Taiwan University Hospital for surgery (radical resection of kidney and ureter or bladder removal) of urothelial carcinoma histopathology specimens of patients willing to participate in this study and the subjects described in the consent Book signer.

Exclusion Criteria:

* In January 2008 to December 2012 at the National Taiwan University Hospital for surgery (radical resection of kidney and ureter or bladder removal) of urothelial carcinoma histopathology specimens of patients are reluctant to join the researcher

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with age between 20-80 years old and had taken Radical Cystectomy or nephrectomy between 2008-2012 were chosen as study population
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The IHC staining score | at the time of surgery
  the IHC staining scores are acquired by IHC staining and assessed by pathologist. The comparisons between each specimen are determined by IHC scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-How Huang, M.D.,Ph.D., Principal Investigator — No. 7, Chung Shans. Rd., Taipei, Taiwan
Locations (2):
- Taiwan (2):
  - Department of Urology, National Taiwan University Hospital, Taipei, No. 7, Chung Shans. Rd.,
  - Department of Urology, National Taiwan University Hospital, Taipei, No. 7, Chung Shans. Rd.

REFERENCES:
- [Background] Hussain SA, James ND. The systemic treatment of advanced and metastatic bladder cancer. Lancet Oncol. 2003 Aug;4(8):489-97. doi: 10.1016/s1470-2045(03)01168-9. PMID 12901963
- [Background] Ueki O, Hisazumi H, Uchibayashi T, Naito K, Tajiri S, Takemae K, Kawaguchi K, Kameda K, Nishino A, Nango C, et al. Methotrexate, vinblastine, doxorubicin, and cisplatin for advanced urothelial cancer. Cancer Chemother Pharmacol. 1992;30 Suppl:S72-6. doi: 10.1007/BF00686947. PMID 1394823
- [Background] Tachibana H. Molecular basis for cancer chemoprevention by green tea polyphenol EGCG. Forum Nutr. 2009;61:156-169. doi: 10.1159/000212748. Epub 2009 Apr 7. PMID 19367120
- [Background] Yang CS, Wang X, Lu G, Picinich SC. Cancer prevention by tea: animal studies, molecular mechanisms and human relevance. Nat Rev Cancer. 2009 Jun;9(6):429-39. doi: 10.1038/nrc2641. PMID 19472429
- [Background] Manning BD, Cantley LC. AKT/PKB signaling: navigating downstream. Cell. 2007 Jun 29;129(7):1261-74. doi: 10.1016/j.cell.2007.06.009. PMID 17604717